CLINICAL TRIAL: NCT06419738
Title: Clinical, Psychosocial, Behavioral Characteristics and Treatment Effectiveness of Low Level Laser Therapy on Patients With Temporomandibular Joint Disorders
Brief Title: Efficacy of Combining Low-Level Laser Therapy With a Self-Management Program on Myalgia in Temporomandibular Disorders
Acronym: LASER-SM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Responsible Party: Principal Investigator, Nguyen Ngoc Hoa, Lecturer, Hanoi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCS01050122107
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Temporomandibular Joint Disorders; Facial Pain
Keywords: temporomandibular joint disorders, temporomandibular disorders, low-level laser therapy, temporomandibular disorders treatment; temporomandibular joint disorders; temporomandibular disorders; low-level laser therapy; self - management program; occlusal splint; Treatment of temporomandibular disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders; Facial Pain | interventions — Self-Management

STUDY DESIGN:
Intervention Model Description: 66 patients were divided into 3 groups.Patients without treatment (because of economic or geographical conditions) were persuaded to join the control group. Group 3 includes 22 patients who will be counseled on changing habits, adjusting behavior, exercising and will be taken in order of examination. 44 patients will be randomized into the remaining 2 groups by using Excel software to create a random number table, patients will draw even numbers into group 2, odd numbers into group 1.
  * Group 1: wear stabilization splint at night for 2 months combined with counseling, behavior modification, and exercise.
  * Group 2: recieve low level laser treatment 3 times aweek, 20 seconds each time, 10 times in total, combined with counseling, behavior modification, and exercise.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-Management Program (Active Comparator): Self-Management Program includes education about the disorder, proprioceptive awareness, and reversing parafunctional habits, relaxation techniques, and stress management. Furthermore, patients are also consulted on changing habits, adjusting behavior, and exercising. Patients are instructed to adjust their behavior: quit harmful habits to limit pain in daily functional activities, maintain scientific sleep, maintain good head, neck, and shoulder activities, soft diet and avoid hard foods, do exercises twice a day: open mouth wide combined with cool compresses and warm compresses.
  Interventions: Behavioral: Self-Management Program
- Low level laser therapy combined with Self-Management Program (Experimental): LLLT may facilitate the release of endogenous opioids, tissue repairment and cellular respiration, increase vasodilatation and pain threshold, and decrease inflammation. Diode low-energy laser machine (Sirolaser blue, Dentsply) are set the default mode according to the correct parameters before use: wavelength 660nm, energy level 2.5 J/cm2, power source 100mW. The projection head is placed perpendicular to the muscle being projected. The laser light is shone on the pain point at the beginning of the treatment, then it will shine on muscle points in turn: temporal muscle (anterior, middle, posterior), masseter muscle (upper, middle, lower), 5 points around the temporomandibular joint area (superior, anterior, lateral, posterior, posterior subcondylar). Each masticatory muscle area is treated for 20 seconds, 3 sessions /week (different days), 10 sessions total. In addition, patients are still instructed Self-Management Program as group 1.
  Interventions: Behavioral: Self-Management Program; Radiation: Low level laser therapy combined with Self-Management Program
- Occlusal Splint combined with Self-Management Program (Active Comparator): Maxillary occlusal splints are made of hard acrylic after taking impressions of the upper dental arches, recording of centric relation (Okeson). Splints are adjusted to provide even occlusal contact during jaw closing and chewing, and canine and incisor contact during protrusive movements of the jaw. Patients are instructed to use the splint each night at least 8 hours/day for a period of 8 weeks. In addition, patients are still instructed Self-Management Program as group 1.
  Interventions: Behavioral: Self-Management Program; Device: Occlusal Splint combined with Self-Management Program

INTERVENTIONS:
Behavioral: Self-Management Program — Self-Management Program includes education about the disorder, proprioceptive awareness and reversing parafunctional habits, relaxation techniques, and stress management. Furthermore, patients are also consulted on changing habits, adjusting behavior, and exercising. Patients are instructed to adjust their behavior: quit harmful habits to limit pain in daily functional activities, maintain scientific sleep, maintain good head, neck, and shoulder activities, soft diet and avoid hard foods, do exercises twice a day: open mouth wide combined with cool compresses and warm compresses.
Radiation: Low level laser therapy combined with Self-Management Program — LLLT may facilitate the release of endogenous opioids, tissue repairment and cellular respiration, increase vasodilatation and pain threshold, and decrease inflammation. Diode low-energy laser machine (Sirolaser blue, Dentsply) are set the default mode according to the correct parameters before use: wavelength 660nm, energy level 2.5 J/cm2, power source 100mW. The projection head is placed perpendicular to the muscle being projected. The laser light is shined on the pain point at the beginning of the treatment, then it will shine on muscle points in turn: temporal muscle (anterior, middle, posterior), masseter muscle (upper, middle, lower), 5 points around the temporomandibular joint area (superior, anterior, lateral, posterior, posterior subcondylar). Each masticatory muscle area is treated for 20 seconds, 3 sessions /week (different days), 10 sessions total. In addition, patients are still instructed Self-Management Program as group 1.
  Arms: Low level laser therapy combined with Self-Management Program
Device: Occlusal Splint combined with Self-Management Program — Maxillary occlusal splints are made of hard acrylic after taking impressions of the upper dental arches, recording of centric relation (Okeson). Splints are adjusted to provide even occlusal contact during jaw closing and chewing, and canine and incisor contact during protrusive movements of the jaw. Patients are instructed to use the splint each night at least 8 hours/day for a period of 8 weeks.In addition, patients are still instructed Self-Management Program as group 1.
  Arms: Occlusal Splint combined with Self-Management Program

SUMMARY:
The purpose of this study is to evaluate the efficacy of combining low-level laser therapy and the self-management program for patients with temporomandibular joint disorders using a randomized controlled design.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of combining low level laser therapy and self-management program for patients with temporomandibular joint disorders using a randomized controlled design.

66 patients suffering from acute and subacute myalgia diagnosed using Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) at High-tech Center for Odonto-Stomatology, Institute of Odonto-Stomatology, Ha Noi Medical University, Viet Nam. Patients without treatment (because of economic or geographical conditions) were persuaded to join the control group. Group 3 includes 22 patients who will be counseled on changing habits, adjusting behavior, exercising and will be taken in order of examination. 44 patients will be randomized into the remaining 2 groups:

* Group 1: wear stabilization splint at night for 2 months combined with counseling, behavior modification, and exercise.
* Group 2: recieve low level laser treatment 3 times aweek, 20 seconds/ session, 10 sessions in total, combined with counseling, behavior modification, and exercise.

Assessment takes place at baseline, after treatment approximately 2 weeks, 4 weeks, 12 weeks, 24 weeks later and 48 weeks follow up. The effects of the interventions are evaluated in terms of reduction in pain intensity (Visual Analogue Scale-VAS), number of masticatory muscle pain point with palpation, number of supplemental muscle pain with palpation, maximum mouth opening, right lateral movements, left lateral movements, protrusive movements, Jaw functional limitation scale (JFLS-8), psychological variables such as PHQ-9, PHQ-4, GAD-7.

Data were entered and analyzed by SPSS 16.0 software. Use Mann-Whitney U test, Kruskal-Wallis test, and Wilcoxon test applied to non-normally distributed variables to compare VAS between groups at different follow-up times. Use paired t-test and independent t-test to compare the maximum opening, lateral movements, protrusive movements, JFLS-8, PHQ-9, PHQ-4, GAD-7 between groups before and after treatment. p value < 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Temporomandibular joint Disorders (according to DC/TMD) with acute or subacute temporal muscle and/or masseter muscle pain (less than 3 months).
* All patients aged 16 years or older, capable of comprehending the doctor's opinion and complying with the examination process.

Exclusion Criteria:

* Patients with chronic TMDs pain, swelling and pain in the mouth that prevent wearing a occlusal splint.
* Patients with history of severe neurological disorders, autoimmune joint and muscle diseases, advanced malignant cancer, history of mental illness, history of alcoholism, drug and painkiller abuse, undergoing surgery and/or radiotherapy on the neck and face, other treatments on the neck and temporomandibular joint within 3 months, use of drugs that may affect the neuromuscular system.
* Pregnant patients

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
VAS | Repeated-measures design with six assessment time points: baseline (pre-treatment), and follow-ups at 2, 4, 12, 24, and 48 weeks.
  The VAS (Visual Analog Scale) pain scale consists of a 10 cm long straight line (without marks), with "no pain" written at the left end and "unbearable pain" written at the right end. Patients were instructed to mark a vertical line above the horizontal line indicating the intensity of their pain. The distance from the zero point to the marker is then measured in millimeters by a caliper. Add the total score of the answers to evaluate the severity according to the following scale: ≤3.4: mild; 3.5-7.4: average; ≥ 7.5: severe
Numbers of masticatory muscle pain with palpation | Repeated-measures design with six assessment time points: baseline (pre-treatment), and follow-ups at 2, 4, 12, 24, and 48 weeks.
  Numbers of muscle pain points are determined by the examiner using a fingertip force of 1kg to palpate the masticatory muscles: temporal muscles (anterior, middle, posterior), masseter muscles (origin, body, attachment, surrounding muscles. Before palpating , the fingertip force needs to be calibrated 3 times with a micro scale, touching each side one by one.
Maximum mouth opening | Repeated-measures design with six assessment time points: baseline (pre-treatment), and follow-ups at 2, 4, 12, 24, and 48 weeks.
  Maximum mouth opening (MMO) was defined asthe maximal interincisal distance on unassisted active mouth opening when the patient opens his mouth maximally without feeling pain. Use a ruler with mm value.
Numbers of supplemental muscle pain with palpation | Repeated-measures design with six assessment time points: baseline (pre-treatment), and follow-ups at 2, 4, 12, 24, and 48 weeks.
  Numbers of supplemental muscle pain points are determined by the examiner using a fingertip force of 1kg to palpate the masticatory muscles: temporal muscles (anterior, middle, posterior), masseter muscles (origin, body, attachment, surrounding muscles. Before palpating , the fingertip force needs to be calibrated 3 times with a micro scale, touching each side one by one.

SECONDARY OUTCOMES:
Right lateral movements | Repeated-measures design with six assessment time points: baseline (pre-treatment), and follow-ups at 2, 4, 12, 24, and 48 weeks.
  Ask the patient to open slightly, and to move his or her jaw as far as he/she can to the right, even if it is painful. Measure from the maxillary reference midline to the mandibular reference midline.
Left lateral movements | Repeated-measures design with six assessment time points: baseline (pre-treatment), and follow-ups at 2, 4, 12, 24, and 48 weeks.
  Ask the patient to open slightly, and to move his or her jaw as far as he/she can to the left, even if it is painful. Measure from the maxillary reference midline to the mandibular reference midline.
Protrusive movements | Repeated-measures design with six assessment time points: baseline (pre-treatment), and follow-ups at 2, 4, 12, 24, and 48 weeks.
  Ask the patient to open slightly, and to move his or her jaw as far as he/she can forward, even if it is painful. Measure the distance from the buccal surface of the mandibular tooth to the buccal surface of the maxillary tooth.
JFLS-8 | Repeated-measures design with six assessment time points: baseline (pre-treatment), and follow-ups at 2, 4, 12, 24, and 48 weeks.
  JFLS-8 (Jaw Functional Limitation Scale - 8) according to DC/TMD axis II to evaluate the level of mandibular function limitation in the past 30 days. The patient will be instructed to answer the questionnaire: in case the patient avoids the activity completely because it is too difficult to do, the patient will circle '10'. If the patient avoids an activity not for pain or difficulty, he/ she will leave this section blank. Activities include: chewing hard foods, chewing chicken, eating soft foods without chewing, opening mouth wide enough to drink from a cup, swallowing, yawning, speaking, laughing.
GAD-7 | Repeated-measures design with six assessment time points: baseline (pre-treatment), and follow-ups at 2, 4, 12, 24, and 48 weeks.
  General anxiety symptoms were assessed using the 7-item scale from the Patient Health Questionnaire (GAD-7). The GAD-7 asks for anxiety symptoms during the past month on a 1 ('not at all') to 3 ('more than half of the days') rating scale (range 7-21). Higher scores indicate higher levels of anxiety.
PHQ-9 | Repeated-measures design with six assessment time points: baseline (pre-treatment), and follow-ups at 2, 4, 12, 24, and 48 weeks.
  Patient Health Questionnaire-9 is a depression assessment form. Patients answer questions consisting of 9 items. Responses will be scored as follows: none: 0 points; several days: 1 point; more than half of the days of the week: 2 points; almost every day: 3 points. Add the total score of the answers to evaluate the severity according to the following scale: 0-4 points: normal; 5-9 points: mild; 10-14 points: average; 15-19 points: quite severe; 20-27 points: severe.
OBC | Repeated-measures design with six assessment time points: baseline (pre-treatment), and follow-ups at 2, 4, 12, 24, and 48 weeks.
  Oral behaviors checklist (OBC) is to determine the presence of parafunctional behaviors. The score is calculated by summing the validation scores of the corresponding items. Response options are scored 0-4 for each item. Based on a comparison of people with chronic TMDs to people without TMDs, scores of 0-16 are normal, while scores of 17-24 occur twice as often in people with TMDs, and scores of 25-62 occur 17 times more often. Acting as a risk factor for TMDs, a score between 25-62 contributes to the onset of TMDs

CONTACTS AND LOCATIONS:
Locations (1):
- High-tech center for Ondonto-stomatology, Institute of Odonto-Stomatology, Ha Noi Medical University, Hà Nội, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided
Investigators have no plans to publish data related to research participants because all patients included in the doctoral training project of Hanoi Medical University have signed a commitment not to disclose information about the patients in the Ethics Committee's Consent to Participate.

REFERENCES:
- [Result] Ahrari F, Madani AS, Ghafouri ZS, Tuner J. The efficacy of low-level laser therapy for the treatment of myogenous temporomandibular joint disorder. Lasers Med Sci. 2014 Mar;29(2):551-7. doi: 10.1007/s10103-012-1253-6. Epub 2013 Jan 15. PMID 23318917
- [Result] Ahmad SA, Hasan S, Saeed S, Khan A, Khan M. Low-level laser therapy in temporomandibular joint disorders: a systematic review. J Med Life. 2021 Mar-Apr;14(2):148-164. doi: 10.25122/jml-2020-0169. PMID 34104237
- [Result] Xu GZ, Jia J, Jin L, Li JH, Wang ZY, Cao DY. Low-Level Laser Therapy for Temporomandibular Disorders: A Systematic Review with Meta-Analysis. Pain Res Manag. 2018 May 10;2018:4230583. doi: 10.1155/2018/4230583. eCollection 2018. PMID 29861802
- [Result] Ayyildiz S, Emir F, Sahin C. Evaluation of Low-Level Laser Therapy in TMD Patients. Case Rep Dent. 2015;2015:424213. doi: 10.1155/2015/424213. Epub 2015 Oct 26. PMID 26587294
- [Result] Desai AP, Roy SK, Semi RS, Balasundaram T. Efficacy of Low-Level Laser Therapy in Management of Temporomandibular Joint Pain: A Double Blind and Placebo Controlled Trial. J Maxillofac Oral Surg. 2022 Sep;21(3):948-956. doi: 10.1007/s12663-021-01591-4. Epub 2021 May 25. PMID 36274894
- [Result] Basili M, Barlattani A Jr, Venditti A, Bollero P. Low-level laser therapy in the treatment of muscle-skelet pain in patients affected by temporo-mandibular disorders. Oral Implantol (Rome). 2017 Jan 21;10(4):406-411. doi: 10.11138/orl/2017.10.4.406. eCollection 2017 Oct-Dec. PMID 29682258
- [Result] Farshidfar N, Farzinnia G, Samiraninezhad N, Assar S, Firoozi P, Rezazadeh F, Hakimiha N. The Effect of Photobiomodulation on Temporomandibular Pain and Functions in Patients With Temporomandibular Disorders: An Updated Systematic Review of the Current Randomized Controlled Trials. J Lasers Med Sci. 2023 Aug 5;14:e24. doi: 10.34172/jlms.2023.24. eCollection 2023. PMID 37744015
- [Result] Demirkol N, Sari F, Bulbul M, Demirkol M, Simsek I, Usumez A. Effectiveness of occlusal splints and low-level laser therapy on myofascial pain. Lasers Med Sci. 2015 Apr;30(3):1007-12. doi: 10.1007/s10103-014-1522-7. Epub 2014 Feb 7. PMID 24504660
- See also: Efficacy of Low-Level Laser Therapy in Management of Temporomandibular Joint Pain: A Double Blind and Placebo Controlled Trial — https://link.springer.com/10.1007/s12663-021-01591-4